CLINICAL TRIAL: NCT00484887
Title: Characterization of Explanted Hernia Meshes From Human Subjects: A Multi-Center, Prospective Study
Status: Terminated | Type: Observational
Why Stopped: PI left institution
Sponsor: University of Missouri-Columbia (Other)
Collaborators: Mayo Clinic (Other); Washington University School of Medicine (Other); University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: MO-5006-1076737
Record Dates: First submitted 2007-06-07; First posted 2007-06-11 (Estimated); Last update posted 2016-08-08 (Estimated); Status verified 2016-05

CONDITIONS: Pathological Conditions, Signs and Symptoms; Hernia
Keywords: Hernia mesh; Implanted mesh material; Explanted mesh material
MeSH Terms: conditions — Pathological Conditions, Signs and Symptoms; Hernia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Explanted mesh from surgical procedures.
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will collect a large amount of hernia mesh explants and study the changes that occur in the materials in vivo to use the information to help design new mesh made from novel materials. We will have evidence that our current options are not only inadequate but can lead to complications. One of our main goals is to convince our colleagues to change their surgical practice by publishing and educating them with this data.

DETAILED DESCRIPTION:
This study will collect a large amount of hernia mesh explants and study the changes that occur in the materials in vivo to use the information to help design new mesh made from novel materials. We will have evidence that our current options are not only inadequate but can lead to complications. One of our main goals is to convince our colleagues to change their surgical practice by publishing and educating them with this data. The objectives of this study are to establish the largest collection of explanted mesh materials in the country; demonstrate by common testing utilized by materials engineers, that in vivo exposure of mesh to the oxidants produced by phagocytosis may lead to chain scission, production of free radicals, and overall degradation of the material both physically and chemically; test mesh materials for a decrease in compliance, which would account for a tendency of mesh to stiffen while in the body reducing abdominal mobility and leading to chronic pain; characterize the histologic reaction of tissues to mesh; and utilize de-identified patient demographics to identify possible clinical characteristics which affect mesh degradation.

ELIGIBILITY:
Inclusion Criteria:

* Adults (persons 18 and older)
* Previous placement of hernia mesh material
* Current need for excision of previous mesh placement or current need for intra-abdominal surgical procedure

Exclusion Criteria:

* No retained mesh prosthetic
* Non surgical candidate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Surgical patients at the University of Missouri Healthcare system.
Sampling Method: Non-Probability Sample
Enrollment: 272 (Actual)
Dates: Start 2007-04; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Ramshaw, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri Hospital and Clinics, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No